CLINICAL TRIAL: NCT02043314
Title: New Strategy for Treating Latent Tuberculosis Infection in Brazil: A Bioequivalence Study of Two Different Dosages of Isoniazid Tablet Formulations in Human Healthy Volunteers
Brief Title: A Bioequivalence Study of Two Different Dosages of Isoniazid Tablet Formulations in Human Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 03.ISZ18-08BE.02
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoniazida-LAQFA® (Active Comparator): 3 coated tablet of 100mg
  Interventions: Drug: Isoniazida
- Isoniazida (Experimental): coated tablet of 300mg
  Interventions: Drug: Isoniazida

INTERVENTIONS:
Drug: Isoniazida

SUMMARY:
The recommended treatment for latent tuberculosis infection for adults is a daily dose of isoniazid 300mg during 6 months. In Brazil, isoniazid was formulated as 100 mg tables. The treatment duration and the high pill burden compromised patient adherence to the treatment. The Brazilian National Programme for Tuberculosis requested the development of a new 300mg isoniazid formulation. The aim of the study is to compare the bioavailability of the isoniazid 300mg new formulation and three 100mg tablets of the reference formulation.

The study is a randomized, single dose, open label, fasting, two-phase crossover bioequivalence study with a wash out period of 7 days (>7 half-life) in 28 healthy human volunteers. For the determination of isoniazid in human plasma, the investigators developed and validated a sensitive, simple and rapid HPLC-MS/MS method.

This will support the strategy adopted by the Brazilian National Program for Tuberculosis for the treatment of latent tuberculosis. The new formulation will increase patients' adherence to the treatment and quality of life. Medical doctors in Brazil should become aware of the new formulation and the new treatment strategy in order to prescribe the right medication and avoid errors that could result in a high frequency of adverse events. Future research studies should evaluate pharmacovigilance, acceptability of the new tablet formulation and its impact on the cure rate.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* aged between 18 and 50 years
* BMI between 18.5 and 29.9 kg/m²

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Average bioequivalence based on the 90% CI | up to 6 months
  The 90% confidence interval for isoniazid log transformed Cmax and AUC0-t should be within the accepted bioequivalence range 80.00-125.00% for Cmax and AUC0-t of isoniazid.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo W Barroso, Dr, Principal Investigator — Fundação Oswaldo Cruz
Locations (1):
- Synchrophar - Ass. e Desenv. de Projetos Clínicos Ltda., Campinas, São Paulo, Brazil